CLINICAL TRIAL: NCT00801723
Title: Randomised, Double-Blind, Multi-Centre, 12 Month Extension Study to Evaluate the Safety And Efficacy of Daily Budesonide MMX 6 mg Versus Placebo in the Maintenance of Remission in Subjects With Ulcerative Colitis.
Brief Title: (CB-01-02/04) Extension Study of Budesonide Multi-Matrix System (MMX) 6 mg in Maintenance Of Remission In Patients With Ulcerative Colitis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CB-01-02/04
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Results first posted 2020-08-17 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: Budesonide MMX® 6 mg (Experimental): One Budesonide-MMX® 6 mg tablet self-administered by the patients with a glass of water, in the morning after breakfast.
  Interventions: Drug: Budesonide MMX 6 mg Tablet
- 2: Placebo (Placebo Comparator): One placebo tablet self-administered by the patients with a glass of water, in the morning after breakfast.
  Interventions: Drug: Placebo Tablet

INTERVENTIONS:
Drug: Budesonide MMX 6 mg Tablet — Budesonide MMX 6 mg Tablet once daily.
  Arms: 1: Budesonide MMX® 6 mg
Drug: Placebo Tablet — Placebo Tablet once daily.
  Arms: 2: Placebo

SUMMARY:
Randomized, double-blind, comparative study versus placebo performed in patients from studies CB-01-02/01 (NCT00679432), CB-01-02/02 (NCT00679380), or CB-01-02/06 (NCT01100112) who achieved ulcerative colitis disease activity index (UCDAI) remission after 8 weeks of treatment.

Patients in remission at the End of Study visit will be given the opportunity to enter the 12-month Maintenance Phase study outlined in this protocol (CB-01-02/04). The End of Study visit in studies 01, 02, and 06 will be set as the Visit 1 (Day 0) of this study. There will be no interruption of study treatment between the parent studies and this study.

It is planned that approximately 150 patients will be enrolled in the study. Patients will be randomly assigned to two groups to receive either budesonide MMX 6 mg or placebo irrespective of the treatment assigned in studies 01, 02, or 06. Treatments will be administered once a day after breakfast for a maximum of 12 months or up to the occurrence of the first clinical relapse, where clinical relapse is defined as combined recurrence of rectal bleeding and stool frequency ≥ 1-2 stools/day above normal for the patient (score ≥ 1 in both UCDAI items).

During the study, patients will be assessed for safety and efficacy at Visit 1 and after 1, 3, 6, 9, and 12 months of treatment.

Patients will be contacted by telephone on a monthly basis for safety assessment. In case of occurrence of symptoms suggestive of clinical relapse, patients will attend an unscheduled visit at any time during the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling the following criteria are eligible for participation in the study:

  * Male and female patients, 18-75 years old, who are able to understand and voluntarily provide written informed consent.
  * Patients in UCDAI remission defined as a UCDAI score ≤ 1 point with a score of 0 for rectal bleeding and stool frequency, and a ≥ 1 point reduction from baseline in the endoscopy score without any sign of mucosal friability (score 0 for mucosal appearance).
  * Patients who have completed all End of Study assessments for the CB-01-02/01, CB-01-02/02 and CB-01-02/06 studies.
  * Females of child-bearing potential must have had a serum pregnancy test performed at the End of Study visit of the parent studies and must use an acceptable contraceptive method throughout the study treatment period.

Exclusion Criteria:

* Patients who meet any of the following criteria at screening visit are to be excluded from study participation:

  * Subjects who have withdrawn from studies CB-01-02/01, CB 01 02/02 or CB-01-02/06.
  * Subjects who did not achieve induction of remission according to the primary endpoint definition in studies CB-01-02/01, CB 01 02/02 or CB-01-02/06 (i.e. clinical remission defined as a UCDAI score ≤ 1 point with a score of 0 for rectal bleeding and stool frequency, and ≥ 1 point reduction from baseline in the endoscopy score without any sign of mucosal friability [score 0 for mucosal appearance]).
  * Subjects with bone density lower than normal by age and sex (T-score lower than -1) as assessed via dual energy X-ray absorptiometry (DXA) scans.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2008-12; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Eric Sands, Principal Investigator — Massachusetts General Hospital; Simon Travis, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (58):
- United States (53):
  - Santarus Clinical Investigational Site 5051, Huntsville, Alabama
  - Santarus Clinical Investigational Site 5088, Tucson, Arizona
  - Santarus Clinical Investigational Site 5044, Anaheim, California
  - Santarus Clinical Investigational Site 5087, Lakewood, California
  - Santarus Clinical Investigational Site 5033, Los Angeles, California
  - Santarus Clinical Investigational Site 5070, Palm Springs, California
  - Santarus Clinical Investigational Site 5067, San Diego, California
  - Santarus Clinical Investigational Site 5064, Lakewood, Colorado
  - Santarus Clinical Investigational Site 5089, Boynton Beach, Florida
  - Santarus Clinical Investigational Site 5041, Hollywood, Florida
  - Santarus Clinical Investigational Site 5055, New Smyrna Beach, Florida
  - Santarus Clinical Investigational Site 5074, Port Orange, Florida
  - Santarus Clinical Investigational Site 5032, Tampa, Florida
  - Santarus Clinical Investigational Site 5009, Tampa, Florida
  - Santarus Clinical Investigational Site 5047, Winter Park, Florida
  - Santarus Clinical Investigational Site 5003, Zephyrhills, Florida
  - Santarus Clinical Investigational Site 5016, Atlanta, Georgia
  - Santarus Clinical Investigational Site 5056, Columbus, Georgia
  - Santarus Clinical Investigational Site 5068, Evanston, Illinois
  - Santarus Clinical Investigational Site 5008, Metairie, Louisiana
  - Santarus Clinical Investigational Site 5090, Annapolis, Maryland
  - Santarus Clinical Investigational Site 5025, Baltimore, Maryland
  - Santarus Clinical Investigational Site 5092, Hollywood, Maryland
  - Santarus Clinical Investigational Site 5077, Prince Frederick, Maryland
  - Santarus Clinical Investigational Site 5010, Chesterfield, Michigan
  - Santarus Clinical Investigational Site 5006, Troy, Michigan
  - Santarus Clinical Investigational Site 5004, Wyoming, Michigan
  - Santarus Clinical Investigational Site 5005, Marlton, New Jersey
  - Santarus Clinical Investigational Site 5011, Great Neck, New York
  - Santarus Clinical Investigational Site 5101, New York, New York
  - Santarus Clinical Investigational Site 5020, Pittsford, New York
  - Santarus Clinical Investigational Site 5096, Fayetteville, North Carolina
  - Santarus Clinical Investigational Site 5058, Huntersville, North Carolina
  - Santarus Clinical Investigational Site 5091, New Bern, North Carolina
  - Santarus Clinical Investigational Site 5045, Cincinnati, Ohio
  - Santarus Clinical Investigational Site 5078, Dayton, Ohio
  - Santarus Clinical Investigational Site 5001, Yukon, Oklahoma
  - Santarus Clinical Investigational Site 5066, Duncansville, Pennsylvania
  - Santarus Clinical Investigational Site 5065, Pottstown, Pennsylvania
  - Santarus Clinical Investigational Site 5035, Sayre, Pennsylvania
  - Santarus Clinical Investigational Site 5021, Austin, Texas
  - Santarus Clinical Investigational Site 5076, Houston, Texas
  - Santarus Clinical Investigational Site 5019, Houston, Texas
  - Santarus Clinical Investigational Site 5036, Houston, Texas
  - Santarus Clinical Investigational Site 5063, Irving, Texas
  - Santarus Clinical Investigational Site 5072, Kingwood, Texas
  - Santarus Clinical Investigational Site 5054, La Porte, Texas
  - Santarus Clinical Investigational Site 5030, Lewisville, Texas
  - Santarus Clinical Investigational Site 5093, Plano, Texas
  - Santarus Clinical Investigational Site 5100, San Antonio, Texas
  - Santarus Clinical Investigational Site 5079, San Antonio, Texas
  - Santarus Clinical Investigational Site 5015, Salt Lake City, Utah
  - Santarus Clinical Investigational Site 5097, Christiansburg, Virginia
- Canada (5):
  - Santarus Clinical Investigational Site 6014, Vancouver, British Columbia
  - Santarus Clinical Investigational Site 6008, Victoria, British Columbia
  - Santarus Clinical Investigational Site 6004, Richmond Hill, Ontario
  - Santarus Clinical Investigational Site 6006, Toronto, Ontario
  - Santarus Clinical Investigational Site 6013, Longueuil, Quebec

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 2: Placebo | 1: Budesonide MMX® 6 mg
Started | 61 | 62
Completed | 25 | 27
Not Completed | 36 | 35

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2: Placebo | 1: Budesonide MMX® 6 mg | Total
Number analyzed (Participants) | 61 | 62 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.0 (11.77) | 42.9 (12.65) | 42.5 (12.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 26 | 54
  Male | 33 | 36 | 69

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Clinical Remission
Description: Clinical remission was defined as the combined absence of recurrence of rectal bleeding and absence of increased stool frequency.
Time Frame: 1, 3, 6, 9, and 12 months
Population: Number of participants with sufficient diary data to enable determination of clinical remission status at the indicated visit.
Measure: Number; unit: percentage of participants
Arm/Group | 2: Placebo | 1: Budesonide MMX® 6 mg
Number analyzed (Participants) | 32 | 39
percentage of participants
  1 month | 76.7 | 88.2
  3 months | 92.0 | 96.8
  6 months | 76.2 | 80.0
  9 months | 86.7 | 95.0
  12 months | 84.6 | 93.3

2. Secondary Outcome: Percentage of Participants With Clinical Relapse
Description: Clinical relapse was defined as the recurrence of rectal bleeding and/or an abnormal stool frequency [≥ 1-2 stools/day above normal for the participant. Clinical remission/relapse status was based on participant diary entries prior to each scheduled visit.
Time Frame: 12 months
Population: Participants with sufficient diary data to enable determination of clinical relapse status.
Measure: Count of Participants; unit: Participants
Arm/Group | 2: Placebo | 1: Budesonide MMX® 6 mg
Number analyzed (Participants) | 32 | 39
Participants | 19 | 12

3. Secondary Outcome: Percentage of Participants With Endoscopic Relapse
Description: Endoscopic relapse was defined as an increase of ≥ 2 points in the Endoscopic Index score from the value calculated at baseline. The score is comprised of four components (granulated scattering reflected light, vascular pattern, vulnerability of mucosa, and mucosal damage). Scores range from 0 to 12, and higher scores indicate more severe (worse) endoscopic findings.
Time Frame: 12 months
Population: Participants with sufficient index score data to enable determination of endoscopic relapse status.
Measure: Count of Participants; unit: Participants
Arm/Group | 2: Placebo | 1: Budesonide MMX® 6 mg
Number analyzed (Participants) | 32 | 39
Participants | 16 | 27

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | 2: Placebo | 1: Budesonide MMX® 6 mg
Serious Adverse Events (participants affected / at risk) | 1/61 | 1/62
Other Adverse Events (participants affected / at risk) | 30/61 | 34/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 2: Placebo (N=61) | 1: Budesonide MMX® 6 mg (N=62)
Lobar pneumonia (Infections and infestations) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 2: Placebo (N=61) | 1: Budesonide MMX® 6 mg (N=62)
Colitis ulcerative (Gastrointestinal disorders) | 16 | 11
Abdominal pain (Gastrointestinal disorders) | 5 | 6
Headache (Nervous system disorders) | 2 | 4
Osteopenia (Musculoskeletal and connective tissue disorders) | 5 | 1
Frequent bowel movements (Gastrointestinal disorders) | 1 | 4
Haematochezia (Blood and lymphatic system disorders) | 1 | 4
Constipation (Gastrointestinal disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact sponsor directly for details.